CLINICAL TRIAL: NCT00600938
Title: A Multicenter, Randomized, Open-label Phase II Trial Evaluating Deferasirox Compared With Deferoxamine in Patients With Cardiac Iron Overload Due to Chronic Blood Transfusions
Brief Title: Evaluating Use of Deferasirox as Compared to Deferoxamine in Treating Cardiac Iron Overload
Acronym: CORDELIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2206; 2007-000766-20 (EudraCT Number)
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Transfusional Iron Overload; Transfusional Hemosiderosis
Keywords: iron overload; cardiac iron; haemosiderosis; myocardial T2*; left ventricular ejection fraction; LVEF; cardiac dysfunction; thalassaemia; Diamond Blackfan anemia; DBA; sideroblastic anemia; myelodysplastic syndromes; MDS (low and INT-1 risk as per the IPSS for MDS); liver MRI; deferasirox; deferoxamine; ICL670; DFO; cardiovascular magnetic resonance imaging
MeSH Terms: conditions — Iron Overload; Hemochromatosis; Thalassemia; Anemia, Diamond-Blackfan; Anemia, Sideroblastic; Myelodysplastic Syndromes | interventions — Deferasirox; Deferoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Deferasirox (Experimental): 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day
  Interventions: Drug: Core Study: Deferasirox; Drug: Deferasirox
- Deferasirox Placebo (Active Comparator): 50 mg/kg/day to 60 mg/kg/day infused subcutaneously in 8- to 12-hour intervals administered 5 to 7 days/week
  Interventions: Drug: Core Study: Deferoxamine; Drug: Deferoxamine
- Extension: deferoxamine to deferasirox (Experimental): "DFO to ICL" (patients who switched from DFO to deferasirox in extension)
  Interventions: Drug: Extension: deferoxamine to deferasirox
- Extension: deferasirox to deferoxamine (Experimental): "ICL to DFO" (patients who switched from deferasirox to DFO in extension)
  Interventions: Drug: Extension: deferasirox to deferoxamine

INTERVENTIONS:
Drug: Core Study: Deferasirox — 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day
  Other Names: "ICL to ICL"
  Arms: Deferasirox
Drug: Core Study: Deferoxamine — 50 mg/kg/day to 60 mg/kg/day infused subcutaneously in 8- to 12-hour intervals administered 5 to 7 days/week
  Other Names: "DFO to DFO"
  Arms: Deferasirox Placebo
Drug: Extension: deferoxamine to deferasirox — 40 mg/kg deferasirox once daily administered 30 minutes before taking food.
  Other Names: "DFO to ICL"
  Arms: Extension: deferoxamine to deferasirox
Drug: Extension: deferasirox to deferoxamine — DFO at a target range of 50 mg/kg/day to 60 mg/kg/day via subcutaneous (sc) infusion lasting a period of 8 to 12 hrs administered for 5 to 7 days per week,
  Other Names: "ICL to DFO"
  Arms: Extension: deferasirox to deferoxamine
Drug: Deferasirox
  Arms: Deferasirox
Drug: Deferoxamine
  Arms: Deferasirox Placebo

SUMMARY:
This is a clinical research study in patients who have iron overload in the heart due to chronic blood transfusions.

The study will have 2 treatment groups and will compare the safety and efficacy of chelation therapy with a medicine called deferasirox (ICL670) with another medicine called deferoxamine (DFO). The study is aimed at finding out which of the two medicines is the best for treating iron overload in the heart.

Patients will be treated for 12 months (core study phase). Patients who complete the core study phase will be offered to continue their study treatment in a 12 months extension phase. During the core and extension, the effects of treatment on iron overload in the heart and the liver will be evaluated using specific magnetic resonance imaging (MRI) assessments.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients, aged 10 years and above, with β-thalassemia major or DBA or sideroblastic anemia on chronic transfusion therapy, having given written consent to participate in the study.
* Patients with cardiac iron as measured by a myocardial T2* value that is ≥ 6ms but not ≥ 20 ms.
* Patients with a lifetime history of at least 50 units of red cell transfusions, and must be receiving at least ≥10 units/yr of red blood cells transfusions.
* Patients with a left ventricular ejection fraction (LVEF) ≥ 56 % as determined by cardiovascular magnetic resonance (CMR).
* Patients with liver iron content (LIC) value ≥ 3 mg Fe / g dw, as determined by liver MRI.

Exclusion criteria:

* Patients with clinical symptoms of cardiac dysfunction.
* Patients unable to undergo study assessments including MRI
* Patients participating in another clinical trial or receiving an investigational drug.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2007-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Nanning, Guangxi, China
- Novartis Investigative Site, Limassol, Cyprus
- Egypt (2):
  - Novartis Investigative Site, Al Mansurah
  - Novartis Investigative Site, Cairo
- Italy (2):
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Genova, GE
- Novartis Investigative Site, Hazmiyeh, Lebanon
- Novartis Investigative Site, Taipei, Taiwan, Taiwan
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Adana, Turkey
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Istanbul
- Novartis Investigative Site, Dubai, Dubai, United Arab Emirates
- United Kingdom (3):
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London

REFERENCES:
- [Derived] Pennell DJ, Porter JB, Piga A, Lai YR, El-Beshlawy A, Elalfy M, Yesilipek A, Kilinc Y, Habr D, Musallam KM, Shen J, Aydinok Y; CORDELIA study investigators. Sustained improvements in myocardial T2* over 2 years in severely iron-overloaded patients with beta thalassemia major treated with deferasirox or deferoxamine. Am J Hematol. 2015 Feb;90(2):91-6. doi: 10.1002/ajh.23876. Epub 2014 Nov 19. PMID 25345697
- [Derived] Pennell DJ, Porter JB, Piga A, Lai Y, El-Beshlawy A, Belhoul KM, Elalfy M, Yesilipek A, Kilinc Y, Lawniczek T, Habr D, Weisskopf M, Zhang Y, Aydinok Y; CORDELIA study investigators. A 1-year randomized controlled trial of deferasirox vs deferoxamine for myocardial iron removal in beta-thalassemia major (CORDELIA). Blood. 2014 Mar 6;123(10):1447-54. doi: 10.1182/blood-2013-04-497842. Epub 2014 Jan 2. PMID 24385534

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients randomized to 1 of 2 treatment grps ICL or DFO, 20 mg/kg/day once daily for 2 wks, followed by 30 mg/kg/day od for 1 wk and 40 mg/kg/day od (DFO) target dose of 50 to 60 mg/kg/day 8 to 12 hour for 5 to 7 days/wk. In ext. pts could either stay in the same grp from core or could switch grps: ICL to ICL, DFO to DFO, DFO to ICL and ICL to DFO
Groups:
- Deferasirox (ICL). For Extension Labeled as ICL to ICL: 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day
- Deferoxamine (DFO). For Extension Labeled as DFO to DFO: 50 mg/kg/day to 60 mg/kg/day infused subcutaneously in 8- to 12-hour intervals administered 5 to 7 days/week
- DFO to ICL (Deferoxamine to Deferasirox): DFO to ICL" (patients who switched from DFO to deferasirox in extension)
- ICL to DFO (Deferasirox to Deferoxamine): ICL to DFO" (patients who switched from deferasirox to DFO in extension)
Period: Core Study
Arm/Group | Deferasirox (ICL). For Extension Labeled as ICL to ICL | Deferoxamine (DFO). For Extension Labeled as DFO to DFO | DFO to ICL (Deferoxamine to Deferasirox) | ICL to DFO (Deferasirox to Deferoxamine)
Started | 98 | 99 | 0 | 0
Core Safety Set | 96 | 91 | 0 | 0
Per Protocol Set (PPS) | 91 | 81 | 0 | 0
Completed | 82 | 78 | 0 | 0
Not Completed | 16 | 21 | 0 | 0
Not completed — Abnormal test procedure result(s) | 3 | 2 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 1 | 2 | 0 | 0
Not completed — Patient withdrew consent | 7 | 12 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0
Period: Extension Study
Arm/Group | Deferasirox (ICL). For Extension Labeled as ICL to ICL | Deferoxamine (DFO). For Extension Labeled as DFO to DFO | DFO to ICL (Deferoxamine to Deferasirox) | ICL to DFO (Deferasirox to Deferoxamine)
Started | 74 (Of the 82 patients who completed the ICL core, 74 continued on the ICL ext. phase; 1 went to ICL-DFO) | 29 (Of the 78 patients who completed the DFO core, 29 went on DFO ext. phase; 42 went to the DFO-ICL) | 42 (Of the 78 patients who completed the DFO core, 29 went on DFO ext. phase; 42 went to the DFO-ICL) | 1 (Of the 82 patients who completed the ICL core, 74 continued on the ICL ext. phase; 1 went to ICL-DFO)
Extension Safety Set | 73 (1 patient did not receive drug in the ext. phase but received drug in the core phase) | 29 | 42 | 1
Completed | 65 | 24 | 33 | 0
Not Completed | 9 | 5 | 9 | 1
Not completed — Adverse Event | 1 | 0 | 2 | 0
Not completed — Abnormal test procedure results | 0 | 1 | 1 | 1
Not completed — Unsatisfactory therapeutic effect | 4 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 3 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0
Not completed — Death | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per Protocol Set (PPS): randomized patients who received at least 6 months of study drug, had a T2* value assessed at least 150 days after randomization, and had no major protocol deviations. A total of 25 patients (7 in the deferasirox arm and 18 in the DFO arm) were excluded from PPS
Groups:
- Core: Deferasirox (ICL): 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day
- Core: Deferoxamine (DFO): 50 mg/kg/day to 60 mg/kg/day infused subcutaneously in 8- to 12-hour intervals administered 5 to 7 days/week
- Total: Total of all reporting groups
Arm/Group | Core: Deferasirox (ICL) | Core: Deferoxamine (DFO) | Total
Number analyzed (Participants) | 98 | 99 | 197
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.9 (6.53) | 19.7 (6.32) | 19.8 (6.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 58 | 57 | 115

OUTCOME MEASURES:

1. Primary Outcome: Core Study: Change From Baseline in Myocardial T2* (Magnetic Resonance T2-star (T2*) Technique for the Measurement of Tissue Iron) After 12 Months Treatment
Description: Non- inferiority in efficacy of deferasirox compared to deferoxamine (DFO) in treating cardiac iron overload as measured by T2*. A non-inferiority margin of 0.9 (90%) was applied. Due to limitations in performing heart biopsies, T2* (T2 star), a Magnetic Resonance (MR) relaxation parameter expressed in milliseconds, as is an important tool to noninvasively quantify cardiac iron concentration. Studies have shown that myocardial T2* evaluations may predict cardiac events, e.g., impaired (<56%) left ventricular ejection fraction (LVEF) is prevalent among patients with low T2*: found in 62% of patients with T2*<8 ms; 20% with T2* of 8-12 ms; and in 5% with T2* >12 ms (Tanner 2006)
Time Frame: 12 Month
Population: Per Protocol Set (PPS) consisted of all randomized patients who received at least 6 months of randomized study drug, had a T2* value assessed at least 150 days after randomization, adhered to the major inclusion and none of the major exclusion criteria, and had no major protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: Millisecond
Groups:
- Core: Deferasirox (ICL): 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day for 12 months.
- Core: Deferoxamine (DFO): 50 mg/kg/day to 60 mg/kg/day infused subcutaneously in 8- to 12-hour intervals administered 5 to 7 days/week for 12 months.
Arm/Group | Core: Deferasirox (ICL) | Core: Deferoxamine (DFO)
Number analyzed (Participants) | 91 | 81
Millisecond | 1.12 (3.687) [1.07 to 1.18] | 1.07 (2.931) [1.02 to 1.11]

2. Secondary Outcome: Core Study: Cardiac Function After 12 Months of Treatment With Deferasirox vs. Deferoxamine, by Change in Left Ventricular Ejection Fraction (LVEF)
Description: An absolute change from baseline in LVEF after 12 months treatment with deferasirox and compared to.DFO was tested using an analysis of covariance model including baseline left ventricular ejection fraction (LVEF) as a covariate.
Time Frame: 12 Month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Groups:
- Core: Deferasirox (ICL). For Extension Labeled as ICL to ICL: 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day for 12 month
- Core: Deferoxamine (DFO). For Extension Labeled as DFO to DFO: 50 mg/kg/day to 60 mg/kg/day infused subcutaneously in 8- to 12-hour intervals administered 5 to 7 days/week for 12 month
Arm/Group | Core: Deferasirox (ICL). For Extension Labeled as ICL to ICL | Core: Deferoxamine (DFO). For Extension Labeled as DFO to DFO
Number analyzed (Participants) | 91 | 81
Percent | -0.5 (0.47) [1.07 to 1.18] | -0.0 (0.49) [1.02 to 1.11]

3. Secondary Outcome: Core Study: Cardiac Function After 6 Months of Treatment With Deferasirox vs. Deferoxamine, by Change in Left Ventricular Ejection Fraction (LVEF)
Description: An absolute change from baseline in LVEF after 6 months treatment with deferasirox and DFO was summarized
Time Frame: 6 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Core: Deferasirox (ICL). For Extension Labeled as ICL to ICL | Deferoxamine (DFO). For Extension Labeled as DFO to DFO
Number analyzed (Participants) | 85 | 73
Percent | -0.95 (4.485) | -0.37 (4.389)

4. Secondary Outcome: Core Study: Change From Baseline in Myocardial T2* After 6 Months Treatment
Description: Summary statistics of T2* ratio Month 6/baseline
Time Frame: 6 Month
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Core: Deferasirox (ICL). For Extension Labeled as ICL to ICL | Core: Deferoxamine (DFO). For Extension Labeled as DFO to DFO
Number analyzed (Participants) | 85 | 73
Ratio | 1.04 (4.752) [1.00 to 1.08] | 1.04 (4.417) [1.00 to 1.08]

5. Secondary Outcome: Core Study: Cardiac Function After 6 and 12 Months Treatment With Deferasirox vs. Deferoxamine, by Change in Left Ventricular End Systolic Volume Indices (LVESVI)
Description: An absolute change from baseline in LVESVI after 6 and 12 months treatment with deferasirox and DFO was summarized. Changes in cardiovascular magnetic resonance (CMR) measured left ventricular end systolic after 6 and 12 months treatment. Left ventricular (LV) end-systolic volume indexed to body surface area (ESVI) is a simple yet powerful echocardiographic marker of LV remodeling that can be measured easily. Left ventricular (LV) end-systolic volume (ESV) has been shown to be an important determinant of survival after myocardial infarction (MI)
Time Frame: 6 Month, 12 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Core: Deferasirox (ICL). For Extension Labeled as ICL to ICL | Core: Deferoxamine (DFO). For Extension Labeled as DFO to DFO
Number analyzed (Participants) | 91 | 81
Milliliter
  Change from baseline at 6 Month (n= 85, 73) | 1.8 (8.021) | 0.88 (8.919)
  Change from Baseline at 12 Month/EOS (n= 91, 81) | 1.57 (8.040) | 0.10 (10.387)

6. Secondary Outcome: Core Study: Core Study: Cardiac Function After 6 and 12 Months of Treatment With Deferasirox vs. Deferoxamine, by Change in Left Ventricular End Diastolic Volume Indices (LVEDVI)
Description: An absolute change from baseline in LVEDVI after 6, and 12 months treatment with deferasirox and DFO was summarized
Time Frame: 6 Month, 12 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- Core; Deferasirox (ICL). For Extension Labeled as ICL to ICL: 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day for 12 month
- Core: Deferoxamine (DFO). For Extension Labeled as DFO to DFO: 50 mg/kg/day to 60 mg/kg/day infused subcutaneously in 8- to 12-hour intervals administered 5 to 7 days/week
Arm/Group | Core; Deferasirox (ICL). For Extension Labeled as ICL to ICL | Core: Deferoxamine (DFO). For Extension Labeled as DFO to DFO
Number analyzed (Participants) | 91 | 81
Percent
  Change from Baseline at 6 Month (n= 85, 73) | 1.81 (14.515) | 1.48 (19.188)
  Change from Baseline at 12 Month/EOS (n= 91, 81) | 1.79 (13.122) | 1.10 (20.485)

7. Secondary Outcome: Core Study: Cardiac Function After 6 and 12 Months of Treatment With Deferasirox vs. Deferoxamine, by Change in Left Ventricular Mass Indices (LVMI)
Description: An absolute change from baseline in LVMI after 6, and 12 months treatment with deferasirox and DFO was summarized
Time Frame: 6 Month, 12 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gram/m^2
Arm/Group | Core: Deferasirox (ICL). For Extension Labeled as ICL to ICL | Core: Deferoxamine (DFO). For Extension Labeled as DFO to DFO
Number analyzed (Participants) | 91 | 81
gram/m^2
  Change from Baseline at 6 Month (n= 85, 73) | 1.01 (13.102) | 3.32 (13.585)
  Change from Baseline at 12 Month/EOS (n= 91, 81) | 4.13 (15.055) | 5.25 (14.973)

8. Secondary Outcome: Core Study: Cardiac Function and the Proportion of Patients Dropping Out Due to Cardiac Dysfunction After Treatment With Deferasirox vs. Deferoxamine
Description: The number of patients withdrawn from the study due to LVEF <50%, T2* <6 ms or significant decreases in T2* ≥ 33% from baseline was provided per treatment group.
Time Frame: 12 Month
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Core; Deferoxamine (DFO). For Extension Labeled as DFO to DFO: 50 mg/kg/day to 60 mg/kg/day infused subcutaneously in 8- to 12-hour intervals administered 5 to 7 days/week for 12 month
Arm/Group | Core: Deferasirox (ICL). For Extension Labeled as ICL to ICL | Core; Deferoxamine (DFO). For Extension Labeled as DFO to DFO
Number analyzed (Participants) | 98 | 99
Participants | 3 | 2

9. Secondary Outcome: Core Study: Safety and Tolerability of Deferasirox vs Deferoxamine Over the 12 Months Treatment Period.
Description: Number of patients with adverse events, serious adverse events and death
Time Frame: 12 Month
Population: Safety Set (SS) consisted of all randomized patients who received at least one dose of study drug and had at least one post-baseline safety assessment. Patients were analyzed according to treatment received. Treatment received is defined as first study drug administered
Measure: Number; unit: Participants
Groups:
- Core: Deferasirox (ICL). For Extension Labeled as ICL to ICL: 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day
Arm/Group | Core: Deferasirox (ICL). For Extension Labeled as ICL to ICL | Core: Deferoxamine (DFO). For Extension Labeled as DFO to DFO
Number analyzed (Participants) | 96 | 91
Participants
  At least one AE | 65 | 69
  Serious Adverse Events | 10 | 10
  Death. None were considered related to study drug. | 1 | 1

10. Secondary Outcome: Core Study: Single and Repeated Dose Pharmacokinetics of Deferasirox, Area Under the Plasma Concentration-time Curve for a Dosing Interval (AUCtau)
Description: The plasma level of deferasirox (ICL670) obtained in this study was summarized descriptively. Plasma concentration was plotted by patient and by visit. Descriptive statistics included the mean, median, SD, and CV, min and max. deferasirox pharmacokinetics (PK) trough levels over the 12 months of treatment and obtained PK profiles for the 40 mg/kg/day deferasirox dose, area under the plasma concentration-time curve for a dosing interval (AUCtau)
Time Frame: 12 Month
Population: Pharmacokinetic Analysis Set (PAS): PAS 2: All randomized patients who received the same dose of deferasirox for at least four consecutive days prior to PK sample collection and completed PK sample collection specified in the protocol at Visit 3 or Visit 4 (pre-dose, 1, 2, and 4 hours post-dose).
Measure: Mean (Standard Deviation); unit: (h.ng/mL)
Arm/Group | Deferasirox (ICL). For Extension Labeled as ICL to ICL
Number analyzed (Participants) | 13
(h.ng/mL) | 2129.70 (930.202)

11. Secondary Outcome: Core Study: Single and Repeated Dose Pharmacokinetics of Deferasirox, Maximum Plasma Concentration (Cmax)
Description: The plasma level of deferasirox (ICL670) obtained in this study was summarized descriptively. Plasma concentration was plotted by patient and by visit. Descriptive statistics included the mean, median, SD, and CV, min and max. deferasirox pharmacokinetics (PK) trough levels over the 12 months of treatment and obtained PK profiles for the 40 mg/kg/day deferasirox dose, maximum plasma concentration (Cmax)
Time Frame: 12 Month
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Deferasirox (ICL). For Extension Labeled as ICL to ICL
Number analyzed (Participants) | 13
umol/L | 150.09 (59.143)

12. Secondary Outcome: Core Study: Single and Repeated Dose Pharmacokinetics of Deferasirox, Time Points of Concentration Data
Description: The plasma level of deferasirox (ICL670) obtained in this study was summarized descriptively. Plasma concentration was plotted by patient and by visit. For trough concentration assessments, a 2-mL blood sample was to be taken on arrival at the study site, i.e. prior to the patient receiving the daily deferasirox dose (pre-dose blood sample). A second 2-mL blood sample was to be taken 2 hours later (post-dose sample). At all other visits (Visits 3 - 14), a pre-dose sample was to be taken. For PK profile assessments, 3 blood samples were taken after 1, 2, and 4 hours post-dose in addition to the 2-mL pre-dose
Time Frame: Month 1 and month 2 (pre-dose, 1,2 and 4 hours post-dose)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: (umol/L)
Arm/Group | Deferasirox (ICL). For Extension Labeled as ICL to ICL
Number analyzed (Participants) | 13
(umol/L)
  Month 1, 0 hour (predose) | 32.25 (21.288) [1.0 to 4.0]
  Month 1, 1 hour (post dos) | 96.32 (35.799)
  Month 1, 2 hour (post dose) | 136.47 (51.831)
  Month 1, 4 hour (post dose) | 133.33 (62.815)
  Month 2, 0 hour (predose) | 38.66 (29.887)
  Month 2, 1 hour (post dose) | 119.48 (38.709)
  Month 2, 2 hour (post dose) | 177.19 (55.343)
  Month 2, 4 hour (post dose) | 180.76 (57.877)

13. Secondary Outcome: Extension Study: Change From Baseline in Myocardial T2* After 24 Months Treatment
Description: The measured T2* values, the ratio (post-baseline / baseline T2*) at Month 6, 12, 18 and 24 was summarized for FAS population along with two-sided 95% CIs. The geometric means of the ratio was presented for all treatment groups
Time Frame: Months 6, 12, 18 and 24
Population: Full Analysis Set (FAS): consisted of all patients enrolled in the extension. Patients were analyzed according to the treatment they were assigned to in the beginning of the extension phase.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- Extension : ICL to ICL: Patients from core continued and received same dose 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day
- Extension: DFO to DFO: Patients from core continued and received same 50 mg/kg/day to 60 mg/kg/day infused subcutaneously in 8- to 12-hour intervals administered 5 to 7 days/week
- Extension; DFO to ICL: DFO to ICL" (patients who switched from DFO to deferasirox in extension)
- Extension: ICL to DFO: ICL to DFO" (patients who switched from deferasirox to DFO in extension)
Arm/Group | Extension : ICL to ICL | Extension: DFO to DFO | Extension; DFO to ICL | Extension: ICL to DFO
Number analyzed (Participants) | 74 | 29 | 42 | 1
Ratio
  Month 6 (n=71,26,40,1) | 1.06 (2.763) [1.01 to 1.11] | 1.05 (2.024) [0.98 to 1.12] | 1.03 (2.778) [0.98 to 1.09] | 1.00 (0) [NA to NA] — 95CI is not available for ICL to DFO group as there is only 1 patient.
  Month 12(n=66, 29, 41, 1) | 1.17 (3.654) [1.11 to 1.24] | 1.06 (2.680) [0.97 to 1.15] | 1.07 (3.411) [1.01 to 1.14] | 1.17 (0) [NA to NA] — 95CI is not available for ICL to DFO group as there is only 1 patient.
  Month 18 (n=68, 26, 39, 1) | 1.24 (5.112) [1.16 to 1.34] | 1.18 (3.748) [1.05 to 1.32] | 1.13 (4.376) [1.04 to 1.23] | 1.05 (0) [NA to NA] — 95CI is not available for ICL to DFO group as there is only 1 patient.
  Month 24 (n=63, 25, 33, 1) | 1.38 (5.277) [1.28 to 1.49] | 1.33 (5.821) [1.13 to 1.55] | 1.21 (4.658) [1.09 to 1.34] | 1.11 (0) [NA to NA] — 95CI is not available for ICL to DFO group as there is only 1 patient.

14. Secondary Outcome: Extension Study: Cardiac Function From Baseline to Month 24 by Change in Left Ventricular Ejection Fraction (LVEF)
Description: Cardiac function endpoints (LVEF) obtained by CMR at baseline, Months 6, 12, 18 and 24 were summarized by means of descriptive statistics. These analyses were conducted for the measured values as well as for the absolute changes from baseline
Time Frame: Months 6, 12, 18 and 24
Population: Full Analysis Set (FAS): consisted of all patients enrolled in the extension. Patients were analyzed according to the treatment they were assigned to in the beginning of the extension phase. Cardiac function parameters over time - excluding patients in Egypt sites.
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- Extension: ICL to ICL: Patients from core continued and received same dose 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day
- Extension: DFO to ICL: DFO to ICL" (patients who switched from DFO to deferasirox in extension)
Arm/Group | Extension: ICL to ICL | Extension: DFO to DFO | Extension: DFO to ICL | Extension: ICL to DFO
Number analyzed (Participants) | 74 | 29 | 42 | 1
Percent
  Month 6 (n=71,26,40,1) | -1.1 (4.96) | -1.8 (3.59) | 0.1 (4.60) | -1.0 (0)
  Month 12 (n= 66,29,42,1) | -0.5 (5.02) | 0.3 (5.13) | 0.0 (3.73) | 0 (0)
  Month 18 (n=68,26,39,1 ) | -0.1 (4.84) | -0.8 (5.14) | -1.3 (3.74) | -10.0 (0)
  Month 24 (n= 63,25,33,1) | 0.6 (4.72) | -0.6 (5.02) | 0.2 (4.82) | -18.0 (0)

15. Secondary Outcome: Extension Study: Cardiac Function From Baseline to Month 24 by Change in Left Ventricular End Systolic Volume Indices (LVESVI)
Description: Cardiac function endpoints (LVESVI) obtained by CMR at baseline, Months 6, 12, 18 and 24 were summarized by means of descriptive statistics. These analyses were conducted for the measured values as well as for the absolute changes from baseline
Time Frame: Months 6, 12, 18 and 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/m^2
Groups:
- Extension: ICL to ICL: Patients from core continued and received same 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day
Arm/Group | Extension: ICL to ICL | Extension: DFO to DFO | Extension: DFO to ICL | Extension: ICL to DFO
Number analyzed (Participants) | 74 | 29 | 42 | 1
mL/m^2
  Month 6 (n=69,26,40,1) | 1.7 (7.98) | 3.4 (10.40) | 0 (8.22) | 1 (0)
  Month 12 (n=64,28,40,1 ) | 1.5 (7.42) | -0.8 (9.74) | 0.6 (9.69) | 2 (0)
  Month 18 (n=67,24,35,1 ) | 2.4 (10.58) | 2.8 (11.54) | 4.1 (6.88) | 28.0 (0)
  Month 24 (n=60,23,33,0 ) | 1.6 (10.21) | 4.3 (8.66) | 1.7 (8.56) | NA (NA) — no participant analyzed

16. Secondary Outcome: Extension Study: Cardiac Function From Baseline to Month 24 by Change in Left Ventricular End Diastolic Volume Indices (LVEDVI)
Description: Cardiac function endpoint (LVEDVI ) obtained by CMR at baseline, Months 6, 12, 18 and 24 were summarized by means of descriptive statistics. These analyses were conducted for the measured values as well as for the absolute changes from baseline
Time Frame: Months 6, 12, 18 and 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Extension: ICL to ICL | Extension: DFO to DFO | Extension: DFO to ICL | Extension: ICL to DFO
Number analyzed (Participants) | 74 | 29 | 42 | 1
mL/m^2
  Month 6 (n=69,26,40,1) | 2.0 (14.19) | 3.5 (21.95) | 0.5 (18.77) | 1.0 (0)
  Month 12 (n=64,28,40,1) | 2.0 (13.49) | -0.6 (18.56) | 3.0 (23.06) | 4.0 (0)
  Month 18 (n=67,24,35,1) | 6.5 (17.80) | 4.2 (19.75) | 8.3 (16.08) | 36.0 (0)
  Month 24 (n=60,23,33,0) | 3.4 (21.15) | 9.5 (14.60) | 5.4 (13.97) | NA (NA) — No participant analyzed

17. Secondary Outcome: Extension Study: Cardiac Function From Baseline to Month 24 by Change in Left Ventricular Mass Indices (LVMI)
Description: Cardiac function endpoints (LVMI) obtained by CMR at baseline, Months 6, 12, 18 and 24 were summarized by means of descriptive statistics. These analyses were conducted for the measured values as well as for the absolute changes
Time Frame: Months 6, 12, 18 and 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: gram/m^2
Arm/Group | Extension: ICL to ICL | Extension: DFO to DFO | Extension: DFO to ICL | Extension: ICL to DFO
Number analyzed (Participants) | 74 | 29 | 42 | 1
gram/m^2
  Month 6 (n=69,26,40,1) | 1.4 (12.37) | 1.8 (15.98) | 3.2 (13.38) | -6.0 (0)
  Month 12 (n=64,28,40,1) | 4.2 (13.90) | 9.1 (14.19) | 3.4 (16.54) | 1 (0)
  Month 18 (n=67,24,35,1) | 4.8 (14.37) | -0.1 (16.87) | 4.0 (14.39) | 37.0 (0)
  Month 24 (n=60,23,33,0) | 5.6 (13.00) | 6.7 (14.96) | 10.3 (13.32) | NA (NA) — No participant analyzed

18. Secondary Outcome: Extension Study: The Cardiac Iron Concentration From T2* Values
Description: Cardiac iron concentration (derived from T2* values) at baseline, Months 6, 12, 18 and 24 were summarized by descriptive statistics. The absolute change from baseline at Months 6, 12, 18 and 24 were also summarized by treatment group. Lliver iron concentration is expressed in units (mg of iron / g of liver tissue dry weight (dw)
Time Frame: Months 6, 12, 18 and 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Extension: ICL to ICL | Extension: DFO to DFO | Extension: DFO to ICL | Extension: ICL to DFO
Number analyzed (Participants) | 74 | 26 | 40 | 1
mg Fe/g dw
  Month 6 (n=71,26,40,1) | -0.12 (0.587) | -0.12 (0.539) | -0.08 (0.465) | 0 (0)
  Month 12 (n=66,29,41,1) | -0.38 (0.674) | -0.12 (0.695) | -0.14 (0.490) | -0.77 (0)
  Month 18 (n=68,26,39,1) | -0.47 (0.789) | -0.45 (0.797) | -0.20 (0.607) | -0.24 (0)
  Month 24 (n=63,25,33,1) | -0.70 (0.834) | -0.69 (0.989) | -0.34 (0.863) | -0.52 (0)

19. Secondary Outcome: Extension Study: Change in Liver Iron Concentration (LIC) From Baseline at Month 24
Description: Results of liver iron content (LIC) measurements by MRI was summarized by descriptive statistics. The absolute value and the absolute change from baseline in LIC at Months 6, 12, 18 and 24 were provided by treatment group.
Time Frame: Months 6, 12, 18 and 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Extension: ICL to ICL | Extension: DFO to DFO | Extension: DFO to ICL | Extension: ICL to DFO
Number analyzed (Participants) | 74 | 29 | 42 | 1
mg Fe/g dw
  Month 6 (n=71,26,38,1) | -4.56 (7.467) | -12.66 (7.821) | -6.30 (7.375) | -3.80 (0)
  Month 12 (n=69,29,40,1) | -10.22 (10.674) | -19.44 (11.446) | -7.98 (9.310) | -3.90 (0)
  Month 18 (n=70,23,38,1) | -12.26 (13.938) | -26.09 (13.443) | -10.87 (11.116) | -2.90 (0)
  Month 24 (n=60,24,33,1) | -15.74 (15.205) | -26.02 (14.867) | -10.96 (11.070) | -3.20 (0)

20. Secondary Outcome: Extension Study: Change in Serum Ferritin From Baseline by Month
Description: Serum ferritin values was summarized by descriptive statistics. Absolute value and the absolute change from baseline in serum ferritin by month was provided by treatment group.
Time Frame: Months 6, 12, 18 and 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Extension: ICL to ICL | Extension: DFO to DFO | Extension: DFO to ICL | Extension: ICL to DFO
Number analyzed (Participants) | 74 | 29 | 42 | 1
ug/L
  Month 6 (n=72,28,38,0) | -626.10 (1541.406) | -1307.14 (1520.877) | -1054.87 (1967.651) | NA (NA) — No participants analyzed
  Month 12 (n=70,29,40,1) | -988.46 (2883.416) | -1877.00 (1877.745) | -1223.73 (1808.056) | -498.00 (0)
  Month 18 (n=66,24,39,1) | -1962.14 (2225.438) | -2426.92 (2685.817) | -1494.82 (1511.257) | -1067.00 (0)
  Month 24 (n=59,24,30,0) | -2239.03 (2178.564) | -2724.00 (2693.583) | -1513.23 (2278.144) | NA (NA) — No participants analyzed

21. Secondary Outcome: Core Study: Single and Repeated Dose Pharmacokinetics of Deferasirox, Maximum Plasma Concentration (Tmax)
Description: The plasma level of deferasirox (ICL670) obtained in this study was summarized descriptively. Plasma concentration was plotted by patient and by visit. Descriptive statistics included the mean, median, SD, and CV, min and max. deferasirox pharmacokinetics (PK) trough levels over the 12 months of treatment and obtained PK profiles for the 40 mg/kg/day deferasirox dose, time to reach maximum plasma concentration (Tmax)
Time Frame: 12 Month
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: (h)
Arm/Group | Deferasirox (ICL). For Extension Labeled as ICL to ICL
Number analyzed (Participants) | 13
(h) | 4.00 (930.202) [1.0 to 4.0]

ADVERSE EVENTS:
Description: Core : The safety set consisted of all randomized patients who received at least one dose of study drug and had at least one post-baseline. safety assessment. Extension: one patient assigned to the deferasirox arm died before receiving treatment in the extension phase
Groups:
- Core Phase - ICL670; Extension Phase - ICL to ICL: Patients from core continued and received same 20 mg/kg/day once daily (od) for 2 weeks, followed by 30 mg/kg/day od for 1 week and a subsequent continuation of 40 mg/kg/day
- Core Phase - DFO; Extension Phase - DFO to DFO: Patients from core continued and received same 50 mg/kg/day to 60 mg/kg/day infused subcutaneously in 8- to 12-hour intervals administered 5 to 7 days/week
- Extension Phase - DFO to ICL: DFO to ICL" (patients who switched from DFO to deferasirox in extension)
- Extension Phase - ICL to DFO: ICL to DFO" (patients who switched from deferasirox to DFO in extension)
Arm/Group | Core Phase - ICL670 | Core Phase - DFO | Extension Phase - ICL to ICL | Extension Phase - DFO to DFO | Extension Phase - DFO to ICL | Extension Phase - ICL to DFO
Serious Adverse Events (participants affected / at risk) | 10/96 | 10/91 | 14/73 | 4/29 | 9/42 | 0/1
Other Adverse Events (participants affected / at risk) | 60/96 | 58/91 | 56/73 | 19/29 | 36/42 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Phase - ICL670 (N=96) | Core Phase - DFO (N=91) | Extension Phase - ICL to ICL (N=73) | Extension Phase - DFO to DFO (N=29) | Extension Phase - DFO to ICL (N=42) | Extension Phase - ICL to DFO (N=1)
Hypersplenism (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypogonadism (Endocrine disorders) | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 1 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0
Amoebiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Yersinia infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Calcium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemosiderosis (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Phase - ICL670 (N=96) | Core Phase - DFO (N=91) | Extension Phase - ICL to ICL (N=73) | Extension Phase - DFO to DFO (N=29) | Extension Phase - DFO to ICL (N=42) | Extension Phase - ICL to DFO (N=1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 4 | 1 | 2 | 2 | 0
Hypogonadism (Endocrine disorders) | 2 | 2 | 0 | 0 | 2 | 1
Conjunctivitis (Eye disorders) | 1 | 2 | 4 | 0 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 2 | 7 | 1 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 5 | 6 | 3 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 4 | 10 | 0 | 9 | 1
Nausea (Gastrointestinal disorders) | 6 | 2 | 4 | 1 | 4 | 0
Vomiting (Gastrointestinal disorders) | 6 | 1 | 6 | 0 | 4 | 0
Fatigue (General disorders) | 1 | 2 | 0 | 0 | 3 | 0
Injection site reaction (General disorders) | 0 | 3 | 0 | 0 | 3 | 0
Pyrexia (General disorders) | 5 | 5 | 6 | 3 | 5 | 1
Acute tonsillitis (Infections and infestations) | 1 | 3 | 1 | 1 | 3 | 0
Bronchitis (Infections and infestations) | 1 | 3 | 1 | 0 | 3 | 0
Influenza (Infections and infestations) | 10 | 6 | 11 | 1 | 7 | 0
Nasopharyngitis (Infections and infestations) | 8 | 4 | 12 | 1 | 6 | 0
Otitis media (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 3 | 2 | 4 | 0 | 3 | 0
Tonsillitis (Infections and infestations) | 1 | 2 | 4 | 1 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 8 | 13 | 1 | 9 | 0
Urinary tract infection (Infections and infestations) | 0 | 4 | 1 | 1 | 4 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 3 | 0
Alanine aminotransferase increased (Investigations) | 9 | 5 | 9 | 2 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 3 | 8 | 1 | 2 | 1
Blood creatinine increased (Investigations) | 8 | 2 | 9 | 1 | 3 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1 | 1 | 3 | 0
Platelet count increased (Investigations) | 2 | 5 | 3 | 6 | 0 | 0
Protein urine present (Investigations) | 11 | 8 | 6 | 1 | 7 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1 | 5 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4 | 5 | 2 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4 | 7 | 1 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3 | 1 | 2 | 1
Headache (Nervous system disorders) | 5 | 5 | 7 | 2 | 4 | 0
Depression (Psychiatric disorders) | 2 | 1 | 4 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 5 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 0 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 6 | 0 | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 4 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 3 | 4 | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety